CLINICAL TRIAL: NCT04133805
Title: The Effect of Viscous Dietary Fibers on LDL-cholesterol: A Systematic Review and Meta-analysis of Randomized Controlled Trials
Brief Title: The Effect of Viscous Dietary Fibers on LDL-cholesterol
Status: Unknown | Type: Observational
Last Known Status: Active, not recruiting
Sponsor: Unity Health Toronto (Other)
Responsible Party: Sponsor
Other Study IDs: Viscous fiber on LDL-C
Record Dates: First submitted 2019-06-24; First posted 2019-10-21 (Actual); Last update posted 2019-10-21 (Actual); Status verified 2019-10

CONDITIONS: Cardiovascular Risk Factor; Hypercholesterolemia
Keywords: viscous fiber; barley b-glucan; oat b-glucan; konjac glucomannan; psyllium; guar gum; pectin
MeSH Terms: conditions — Hypercholesterolemia

STUDY DESIGN:
Observational Model: Other | Time Perspective: Other
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

INTERVENTIONS:
Dietary Supplement: viscous fiber — ex. barley b-glucan, oat b-glucan, konjac glucomannan, psyllium, guar gum, and pectin

SUMMARY:
This systematic review and meta-analysis is aimed to assess the effect of commonly consumed viscous fibers on blood lipids including LDL-C, non-HDL-C, and ApoB.

DETAILED DESCRIPTION:
Medline, Embase, CINAHL, and the Cochrane Central databases were searched through May 13, 2019. Three independent reviews extracted data and assessed risk of bias. Randomized controlled trials that assessed the effect of barley b-glucan, oat b-glucan, konjac glucomannan (KJM), psyllium, guar gum, and pectin, with a study duration of ≥ 3 weeks, in adults with or without hypercholesterolemia were included. Data were pooled using the generic inverse variance method with random effects models and expressed as mean differences with 95% confidence intervals. Heterogeneity was assessed by the Cochran Q statistic and quantified by I2 statistic. Overall quality of the evidence was assessed using the GRADE (Grading of Recommendations Assessment, Development, and Evaluation) approach.

ELIGIBILITY:
Inclusion Criteria:

* Must be a randomized controlled clinical trial with either a parallel or cross-over design
* have a treatment period of at least 3 weeks
* Hypercholesterolemic or normocholesterolemic adults, overweight and obese individuals or individuals with diabetes were all acceptable
* Sources from β-glucan oats, β-glucan barley, konjac, psyllium, guar gum, and pectin were accepted
* The amount of soluble fiber must be reported or measured or must be computable.
* Must be appropriately controlled.
* Must measure one of LDL-C, non-HDL-C or ApoB. These lipid measures can be either primary or secondary outcomes.
* Enough information must be provided to calculate the magnitude of effect, i.e. end of treatment measures and/or change from baseline measures

Exclusion Criteria:

* If the study was insufficiently controlled, i.e. the control was another soluble fiber
* If the soluble fiber was a combination supplement or in whole food sources where the amount of soluble fiber could not be isolated
* If the outcome measures did not include LDL-C, non-HDL-C or ApoB
* If the treatment period was less than 3 weeks
* If the study was from a non-adult population
* If the study provided insufficient information to calculate a magnitude of effect
* Secondary information such as reviews, editorials, commentaries, were excluded
* If the dose was less than 0.4g/day

Min Age: 18 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Study Population: Hypercholesterolemic or normocholesterolemic adults, overweight and obese individuals or individuals with diabetes
Sampling Method: Probability Sample
Enrollment: 7845 (Actual)
Dates: Start 2018-09-17 (Actual); Primary Completion 2019-12 (Estimated); Study Completion 2020-01 (Estimated)

PRIMARY OUTCOMES:
LDL-Cholesterol | ≥ 3 weeks

SECONDARY OUTCOMES:
non-HDL-Cholesterol | ≥ 3 weeks
ApoB | ≥ 3 weeks

CONTACTS AND LOCATIONS:
Locations (1):
- Clinical Risk Factor and Modification Centre, Toronto, Ontario, Canada